# STATISTICAL ANALYSIS PLAN

SMART – A prospective, multicenter registry assessing the embolization of neurovascular lesions using the Penumbra SMART COIL® System

Protocol CLP 10023.B

January 11, 2017

# Contents

| 1 | 0 | verview | 3 |
|----|--------|----------------------------------------|----|
| 2 | S | ample Size | 3 |
| 3 | In | iterim Analysis | 4 |
| 4 | Α | nalysis Populations | 4 |
| | 4.1 | Definitions | 4 |
| 5 | S | tatistical Methods | 4 |
| 6 | В | aseline Characteristics | 5 |
| 7 | S | ubject Disposition | 5 |
| 8 | E | ffectiveness Analysis | 5 |
| | 8.1 | Primary Effectiveness Analysis | 5 |
| | 8.2 | Secondary Effectiveness Analysis | 5 |
| 9 | S | ubgroup Analysis | 6 |
| 10 | ) | Safety Analysis | 7 |
| | 10.1 | 1 Primary Safety Analysis | 7 |
| | 10.2 | 2 Analysis of Adverse Events | 7 |
| | 10.3 | 3 Analysis of Deaths | 7 |
| 11 | | Pooling Across Centers | 8 |
| 12 | )<br>- | Lost to Follow-Up and Missing Data | 8 |
| 13 | } | Changes to Planned Analyses | 8 |
| 14 | | Programming Specifications | 8 |
| 15 | ; | References | .0 |
| Ar | nen | ndix: Mock Tables Listings and Figures | 1 |

#### 1 Overview

SMART is a multicenter, single-arm prospective registry. Its primary objective is to acquire postmarket data on the use of the Penumbra SMART COIL® System (Smart) in the treatment of intracranial aneurysms and other malformations.

Approximately 1,000 subjects with intracranial aneurysms or other malformations treated by Smart will be enrolled across up to 100 sites. All subjects will be allocated to treatment with at least 75% Smart, Penumbra Coil 400™ (PC 400), or Penumbra Occlusion Device (POD®) coils as defined by the number of coils implanted.

The primary efficacy endpoint is the rate of retreatment through one year ± 6 months follow-up. The primary safety endpoint is the rate of procedural (within 24 hours of arterial puncture) device-related serious adverse events.

The secondary efficacy endpoints for the registry are the ability to achieve adequate occlusion at immediate post-procedure (Class I or II Raymond-Roy Occlusion Classification for aneurysms) and the number of times re-access with guidewire was required due to catheter kickout while using SMART/POD/PC 400.

This Statistical Analysis Plan (SAP) elaborates on statistical methods outlined in the registry protocol and presents analysis conventions. The SAP will be signed off before database lock.

# 2 Sample Size

The predetermined sample size of approximately n = 1000 subjects allows the primary efficacy and safety endpoints to be estimated with greater than  $\pm$  2% precision: re-treatment at one-year follow-up (95% CI: 6.6% to 10.0%) and procedural device-related serious adverse events (95% CI: 0.93% to 2.5%).

This analysis applies 95% two-sided binomial proportion confidence intervals using normal approximations to the binomial (SAS v 9.4; SAS Institute, Cary, NC).

These estimates assume 8.3% retreatment through one-year follow-up based on the mean rate observed in eight prior studies cited in the protocol, as weighted by their subject sample sizes. A 1.7% rate of procedural device-related serious adverse events is assumed based on data on file at the sponsor.

### 3 Interim Analysis

No interim efficacy analyses are planned for the purpose of terminating the registry early. However, interim analysis may be performed for the purpose of publication of SMART results.

### 4 Analysis Populations

### 4.1 Definitions

The ITT population will consist of all subjects who sign the informed consent and are enrolled in the registry with Smart, PC 400, or POD accounting for 75% or more of the total number of coils implanted. The ITT population will include only the first lesion treated for each subject. Summary statistics will be developed separately for additional lesions.

The PP population will be constructed by excluding subjects who have major protocol violations that impact endpoint evaluations. Subjects will be classified as screen failures if they are not consented or are consented and not enrolled due to failure to implant at least 75% Smart, PC 400, or POD coils or other reasons.

#### **5 Statistical Methods**

For this single-arm registry, results will primarily be presented as descriptive statistics and two-sided 95% confidence intervals.

Baseline, efficacy, and safety variables will be summarized using tables of descriptive statistics for continuous variables (n, mean, median, SD, and range) or frequency counts and percentages for categorical variables.

Confidence intervals will be developed using confidence bounds on the mean or mean change from admission for continuous variables or binomial proportion intervals under a normal approximation to the binomial for categorical variables.

For results developed using data from more than one visit, summaries will be reported for each visit from the full set of observed data available.

Staged procedures are not retreatments for the purposes of running all SMART registry analyses.

#### 6 Baseline Characteristics

Baseline characteristics will be summarized using descriptive statistics for continuous variables or frequency counts and percentages for categorical variables. Two-sided 95% confidence intervals will also be presented.

A summary table will be reported with key baseline characteristics, including subject demographics, admission functional assessments, and lesion evaluation results.

# 7 Subject Disposition

The number of subjects in the following categories will be recorded:

- Enrolled subjects
- Completed and discontinued subjects
- ITT population
- PP population

Frequency counts and percentages will also be tabulated on the reasons for registry discontinuation: adverse events, death, exclusion for medical reasons, exclusion from registry by investigator, LTFU, withdrawal of consent, or other causes.

# 8 Effectiveness Analysis

# 8.1 Primary Effectiveness Analysis

The primary efficacy outcome is the rate of retreatment through one-year follow-up. Frequency counts and percentages will be reported for the subjects who required retreatment. A two-sided 95% binomial proportion confidence interval will be developed for the retreatment rate using a normal approximation to the binomial. All primary and secondary efficacy endpoint analyses will be run on both the intent-to-treat (ITT) population and the per-protocol (PP) population.

# 8.2 Secondary Effectiveness Analysis

Frequency counts and percentages will be reported for the two secondary efficacy outcomes:

Ability to achieve adequate occlusion at immediate post-procedure: Defined as the
proportion of subjects achieving adequate occlusion based on the investigator's
assessment given anatomical and other considerations at immediate post-procedure.

This endpoint applies to the investigator's Yes/No assessment on whether adequate occlusion was achieved and not the Raymond-Roy Occlusion Scale. Frequency counts and percentages will be reported for this proportion. Two-sided 95% binomial proportion confidence intervals will be developed, using a normal approximation to the binomial.

Re-access with guidewire due to catheter kickout: This endpoint applies to catheter kickout while using SMART/PC 400/POD coils and not other adjunctive coils. Frequency counts and percentages will be reported for the proportion of subjects experiencing 0, 1, 2, and ≥ 3 kickout events. Two-sided 95% binomial confidence intervals with a normal approximation to the binomial will be presented for each frequency count.

## 9 Subgroup Analysis

The following subgroup analyses will be performed for the primary and secondary effectiveness and safety endpoints:

- Actual adjunctive treatment used: Balloon, Stent, Other, None
- Age: < 65, ≥ 65
- Aneurysm location: Extradural ICA, ICA, ACA, MCA, Posterior Circulation, Venous Circulation, Other
- Aneurysm size: Small (Up to 10 mm in the largest diameter), Large (> 10 mm to 25 mm in the largest diameter), Giant (> 25 mm in the largest diameter)
- Aneurysm status: Ruptured, Unruptured
- Lesion nature: Aneurysm, Arteriovenous malformation, Fistula, Other
- Lesion treatment technique: Constructive, Deconstructive
- Neck width: Small neck (< 4 mm neck width), Wide neck (≥ 4 mm Neck Width or Dometo-Neck ratio (defined as Dome Width / Neck Width) < 2)</li>
- Vessel treatment at admission: Initial treatment, Retreatment

For re-access with guidewire due to catheter kickout, which is analyzed based on 0, 1, 2, and ≥ 3 kickout events, subgroup analyses will be performed using the Wilcoxon rank-sum test for subgroup variables with two levels and the Kruskal-Wallis test for subgroup variables with more than two levels. For the other three categorical endpoints, subgroup analysis will be performed using Fisher's Exact test.

## 10 Safety Analysis

### 10.1 Primary Safety Analysis

The primary safety endpoint is the proportion of subjects who experience at least one procedural (within 24 hours of arterial puncture) device-related serious adverse event.

Frequency counts and percentages of subjects experiencing a procedural device-related serious adverse event will be provided. A 95% two-sided binomial proportion confidence interval will be reported using a normal approximation to the binomial.

### 10.2 Analysis of Adverse Events

Only adverse events that are related to the procedure or device, unanticipated adverse device effects (UADE), and all serious adverse events (SAE) from consent through registry exit are reportable under the SMART protocol. Reported adverse event data will be presented for each subject, including actions taken, causality (if appropriate), outcome, seriousness, severity, and start and end dates. The onset of adverse events will also be shown relative (in number of days) to the day of treatment. All adverse events will be reported based on the assessment from the clinical study sites.

Rates of device or procedure related adverse events and serious adverse events will be calculated, broken down by category. These reports will count only the most severe adverse event for each subject and only those categories with at least 3% subjects included. Tabulations and descriptive statistics will be produced, including an analysis by time period: (1) intraprocedural or within 24 hours of procedure and (2) after 24 hours post-procedure.

# 10.3 Analysis of Deaths

Survival curves will be produced using the Kaplan-Meier product limit estimator. Survival will be tracked through registry completion at the one-year follow-up visit. In addition, 95% confidence intervals for the Kaplan-Meier survival curves will be computed and plotted at monthly time intervals.

A frequency table will also be presented containing one-year mortality rates, along with 95% two-sided binomial proportion confidence intervals using a normal approximation to the binomial.

## 11 Pooling Across Centers

To assess the validity of data pooling, heterogeneity across sites will be examined using relevant methods, such as ANOVA (continuous variables), contingency tables or binary logistic regression (categorical variables), or Cox proportional hazards (event time variables). Any sites containing fewer than ten subjects will be aggregated in this analysis.

All sites will conduct the registry according to a common protocol. Monitoring efforts will be allocated to assess whether sites are adhering to the protocol in a standardized manner to minimize the presence of heterogeneity across centers.

### 12 Lost to Follow-Up and Missing Data

Missing data are expected to arise on subjects who discontinue the registry early. For sensitivity purposes, the following additional analyses will be conducted on the primary efficacy endpoint:

- Analyze only subjects with complete one-year retreatment rate data
- For those subjects without any observations after treatment, missing one-year retreatment rate data will be imputed from baseline scores and included in an analysis

# 13 Changes to Planned Analyses

All changes to this Statistical Analysis Plan (SAP) will be listed in a revised SAP or in the SMART clinical registry report.

# 14 Programming Specifications

Statistical analyses will be programmed in SAS 9.4 or later (SAS Institute, Cary, NC) and presented in powerpoint, Word, or pdf format depending on whether a presentation or publication is required.

For Word or pdf output, one-inch margins will be used on all sides of the page, and the headers will be as follows. The left header will contain 'Penumbra Inc.' on the top line and 'Protocol CLP 10023' on the second line. The right header will contain pagination in the format 'Page X of Y'. The left footer will contain a statement 'Last run on DDMONYYYY using database version DDMONYYYY and program [program name.sas]'. The right footer will be blank.

Tables, Listings, and Figures will be titled in the format 'Exhibit X.Y: [Name]' on the first line with a subtitle of 'Intent-to-Treat Population' or 'Per-Protocol Population', as applicable, on the second line. The ITT analysis will be numbered 'X.1', and the PP analysis, if available, will be numbered 'X.2', where X denotes the number of the analysis being run. Pagination will reset to 1 for every new analysis, so that the ITT analysis is 'Page 1 of Y' and the PP analysis, if applicable, is 'Page 2 of Y'. A Table of Contents will be presented in the form 'Exhibit X.Y: [Name].......[Page Number]'.

Tables and listings will be presented using left-justified data and a grid border around each cell. The respective column headers in the tables will contain the name of the table, 'All Subjects (N = [number of subjects])', and '95% Cl' unless otherwise specified in the mock TLFs. Column headers for the listings are presented in the shells.

Continuous variables will be presented as mean  $\pm$  SD (min to max) with one decimal place precision, in the format 'X.X  $\pm$  X.X (X.X to X.X)'.

Categorical variables will be presented as percent (frequency/total) for each category with one decimal place precision in the format 'X.X% (n/N)'. Individual categories will be indented four spaces. All categories will be listed out, and categories with zero observations will be reported in the format '0.0% (0/N)'. P-values will be presented to three decimal places.

Missing data will be presented in listings with dots (.) if the variable is continuous or blank cells if the variable is categorical.

The subgroup analysis table will be repeated in the format given in the mock shells for all subgroups and endpoints specified in the SAP section, 'Effectiveness Subgroup Analysis'. The figure 'Kaplan-Meier Estimates of Probability of Death in Subjects' will present a plot of survival curves and confidence intervals at one-month intervals up to one year.

#### 15 References

Agresti (2014). Categorical Data Analysis. John Wiley & Sons: New Jersey.

CLP SMART – A prospective, multicenter registry assessing the embolization of neurovascular lesions using the Penumbra SMART Coil® System. 10023 protocol, revision B, 23AUG2016.

Debrun GM, et al (1998). Selection of cerebral aneurysms for treatment using Guglielmi detachable coils: the preliminary University of Illinois at Chicago experience. *Neurosurgery*, 43(6), 1281-1295.

Hosmer, Lemeshow, and May (2008). *Applied Survival Analysis: Regression Modeling of Time-to-Event Data*. John Wiley & Sons: New Jersey.

# **Appendix: Mock Tables, Listings, and Figures**

#### Part I. Mock Tables

#### **Site Enrollment**

| Site Enrollment | All Subjects (N = N) |
|-----------------|----------------------|
| 99999 | X.X% (n/N) |

**Subject Follow-Up Visits** 

| Subject Follow-Up Visits | All Subjects (N = N) |
|--------------------------|----------------------|
| Admission Evaluation | X.X% (n/N) |
| Follow-Up | X.X% (n/N) |

**Analysis Populations** 

| Analysis Populations | All Subjects (N = N) |
|----------------------------|----------------------|
| Intent-to-Treat Population | X.X% (n/N) |
| Per Protocol Population | X.X% (n/N) |

**Subject Disposition** 

| oubject Disposition | |
|----------------------------------------|----------------------|
| Subject Disposition | All Subjects (N = N) |
| Enrolled Subjects | X.X% (n/N) |
| Completed Subjects | X.X% (n/N) |
| Discontinued Subjects | X.X% (n/N) |
| Adverse Events | X.X% (n/N) |
| Deceased before Completion | X.X% (n/N) |
| Excluded for Medical Reasons | X.X% (n/N) |
| Excluded from Registry by Investigator | X.X% (n/N) |
| Lost to Follow Up | X.X% (n/N) |
| Withdrew Consent | X.X% (n/N) |
| Other | X.X% (n/N) |

**Demographics** 

| Demographics | All Subjects (N = N) | 95% CI |
|--------------|-------------------------------------|--------------|
| Age | $X.X \pm X.X (X.X \text{ to } X.X)$ | (X.X, X.X) |
| Gender: Male | X.X% (n/N) | (X.X%, X.X%) |

**Medical History** 

| Medical History | All Subjects (N = N) | 95% CI |
|---|---|---|
| | | (X.X%, |
| Previous Stroke | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| Headache | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| Migraine | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| Traumatic Brain Injury | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| Myocardial Infarction | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| Hypertension | X.X% (n/N) | X.X%) |
| | N NO ( ( 1) | (X.X%, |
| Thyroid Disorder | X.X% (n/N) | X.X%) |
| D: 1 1 | N NO( / (N) | (X.X%, |
| Diabetes | X.X% (n/N) | X.X%) |
| Other Deat Medical History | V V0/ (= (N1) | (X.X%, |
| Other Past Medical History | X.X% (n/N) | X.X%) |
| Comily I listomy of Anatomyoma or Malformations | V V0/ (m/NI) | (X.X%, |
| Family History of Aneurysms or Malformations | X.X% (n/N) | X.X%) |
| Polycystic Kidney Disease | X.X% (n/N) | (X.X%,<br>X.X%) |
| Folycystic Mulley Disease | X.X /0 (11/1N) | (X.X%, |
| Fibromuscular Dysplasia | X.X% (n/N) | (A.A.%,<br>X.X%) |
| Tibromusodiai Dyspiasia | 73.770 (11/14) | (X.X%, |
| Smoking | X.X% (n/N) | (X.X%) |
| Omorning | 73.7770 (11/14) | (X.X%, |
| Cocaine Use | X.X% (n/N) | X.X%) |

### **Process Times**

| Process Times | All Subjects (N = N) | 95% CI |
|---|---|---|
| | $X.X \pm X.X$ (X.X to | |
| Total Fluoroscopic Time (Minutes) | (X.X) | (X.X, X.X) |
| Time from First Coil Deployed to Last Coil Detached | $X.X \pm X.X$ (X.X to | |
| (Minutes) | (X.X) | (X.X, X.X) |
| | X.X ± X.X (X.X to | |
| Time from Procedure to Retreatment (Days) | (X.X) | (X.X, X.X) |

## **Lesion Evaluation**

| | All Subjects (N = | 25% 21 |
|-------------------------------|-------------------|--------------|
| Lesion Evaluation | N) | 95% CI |
| Lesions Treated | | |
| 1 | X.X% (n/N) | (X.X%, X.X%) |
| 2 | X.X% (n/N) | (X.X%, X.X%) |
| ≥ 3 | X.X% (n/N) | (X.X%, X.X%) |
| Technique: Constructive | X.X% (n/N) | (X.X%, X.X%) |
| Previous Treatment with Coils | X.X% (n/N) | (X.X%, X.X%) |
| Lesion Nature | | |
| Aneurysm | X.X% (n/N) | (X.X%, X.X%) |
| Fistula | X.X% (n/N) | (X.X%, X.X%) |
| Arteriovenous Malformation | X.X% (n/N) | (X.X%, X.X%) |
| Other | X.X% (n/N) | (X.X%, X.X%) |
| Lesion Side | | |
| Right | X.X% (n/N) | (X.X%, X.X%) |
| Left | X.X% (n/N) | (X.X%, X.X%) |
| Midline | X.X% (n/N) | (X.X%, X.X%) |
| Lesion Location | | |
| Extradural ICA | X.X% (n/N) | (X.X%, X.X%) |
| ICA | X.X% (n/N) | (X.X%, X.X%) |
| ACA | X.X% (n/N) | (X.X%, X.X%) |
| MCA | X.X% (n/N) | (X.X%, X.X%) |
| Posterior Circulation | X.X% (n/N) | (X.X%, X.X%) |
| Venous Circulation | X.X% (n/N) | (X.X%, X.X%) |
| Other | X.X% (n/N) | (X.X%, X.X%) |

## **Adjunctive Treatment**

| Adjunctive Treatment | All Subjects (N = N) | 95% CI |
|-----------------------------------|----------------------|--------------|
| Adjunctive Technology Pre-Planned | X.X% (n/N) | (X.X%, X.X%) |
| Stent-Assisted Coiling | X.X% (n/N) | (X.X%, X.X%) |
| Balloon-Assisted Coiling | X.X% (n/N) | (X.X%, X.X%) |
| Other | X.X% (n/N) | (X.X%, X.X%) |
| Adjunctive Technology Used | X.X% (n/N) | (X.X%, X.X%) |
| Stent-Assisted Coiling | X.X% (n/N) | (X.X%, X.X%) |
| Balloon-Assisted Coiling | X.X% (n/N) | (X.X%, X.X%) |
| Other | X.X% (n/N) | (X.X%, X.X%) |

## Modified Rankin Scale

| Modified Rankin Scale | All Subjects (N = N) | 95% CI |
|-----------------------|-------------------------------------|--------------|
| Admission mRS | $X.X \pm X.X (X.X \text{ to } X.X)$ | (X.X, X.X) |
| 0 to 2 | X.X% (n/N) | (X.X%, X.X%) |
| 0 | X.X% (n/N) | (X.X%, X.X%) |
| 1 | X.X% (n/N) | (X.X%, X.X%) |
| 2 | X.X% (n/N) | (X.X%, X.X%) |
| 3 | X.X% (n/N) | (X.X%, X.X%) |
| 4 | X.X% (n/N) | (X.X%, X.X%) |
| 5 | X.X% (n/N) | (X.X%, X.X%) |
| 6 | X.X% (n/N) | (X.X%, X.X%) |
| One-Year mRS | $X.X \pm X.X (X.X \text{ to } X.X)$ | (X.X, X.X) |
| 0 to 2 | X.X% (n/N) | (X.X%, X.X%) |
| 0 | X.X% (n/N) | (X.X%, X.X%) |
| 1 | X.X% (n/N) | (X.X%, X.X%) |
| 2 | X.X% (n/N) | (X.X%, X.X%) |
| 3 | X.X% (n/N) | (X.X%, X.X%) |
| 4 | X.X% (n/N) | (X.X%, X.X%) |
| 5 | X.X% (n/N) | (X.X%, X.X%) |
| 6 | X.X% (n/N) | (X.X%, X.X%) |

Hunt and Hess Grading Scale

| Hunt and Hess Grading Scale | All Subjects (N = N) | 95% CI |
|---|---|---|
| Admission Hunt and Hess | $X.X \pm X.X (X.X \text{ to } X.X)$ | (X.X, X.X) |
| | X.X% (n/N) | (X.X%, X.X%) |
| II | X.X% (n/N) | (X.X%, X.X%) |
| III | X.X% (n/N) | (X.X%, X.X%) |
| IV | X.X% (n/N) | (X.X%, X.X%) |
| V | X.X% (n/N) | (X.X%, X.X%) |

**Primary Effectiveness Analysis** 

| i iiiiai y ziiootivoiiooo / tiiaiyolo | | |
|---------------------------------------|----------------------|--------|
| Primary Effectiveness Analysis | | |
| Primary Endpoint | All Subjects (N = N) | 95% CI |
| | | (X.X%, |
| Retreatment through Follow-Up | X.X% (n/N) | X.X%) |

**Secondary Effectiveness Analysis** 

| Secondary Effectiveness Analysis Secondary Effectiveness Analysis | | |
|---|---|---|
| Secondary Endpoints | All Subjects (N = N) | 95% CI |
| Adequate Occlusion at Immediate Post-Procedure | X.X% (n/N) | (X.X%, X.X%) |
| Raymond Scale Class I | X.X% (n/N) | (X.X%, X.X%) |
| Raymond Scale Class II | X.X% (n/N) | (X.X%, X.X%) |
| Raymond Scale Class III | X.X% (n/N) | (X.X%, X.X%) |
| Re-Access Attempts with Guidewire due to Catheter Kickout (Smart/PC 400/POD) | | |
| 0 | X.X% (n/N) | (X.X%, X.X%) |
| 1 | X.X% (n/N) | (X.X%, X.X%) |
| 2 | X.X% (n/N) | (X.X%, X.X%) |
| ≥ 3 | X.X% (n/N) | (X.X%, X.X%) |
| Additional Analyses | | |
| Re-Access Attempts with Guidewire due to Catheter Kickout (Other Adjunctive Coils) | | |
| 0 | X.X% (n/N) | (X.X%, X.X%) |
| 1 | X.X% (n/N) | (X.X%, X.X%) |
| 2 | X.X% (n/N) | (X.X%, X.X%) |
| ≥ 3 | X.X% (n/N) | (X.X%, X.X%) |
| First Framing Coil Conformed to Lesion Morphology | | |
| Completely Conformed | X.X% (n/N) | (X.X%, X.X%) |
| Partially Conformed | X.X% (n/N) | (X.X%, X.X%) |
| Compartmentalized | X.X% (n/N) | (X.X%, X.X%) |
| N/A | X.X% (n/N) | (X.X%, X.X%) |
| Packing Density | X.X% (n/N) | (X.X%, X.X%) |
| Occlusion at One Year (Aneurysms) | | |
| Class I | X.X% (n/N) | (X.X%, X.X%) |
| Class II | X.X% (n/N) | (X.X%, X.X%) |
| Class III | X.X% (n/N) | (X.X%, X.X%) |
| Occlusion of Lesion at One Year (Non-Aneurysms) | | |
| Better (Progressive Occlusion) | X.X% (n/N) | (X.X%, X.X%) |
| Stable | X.X% (n/N) | (X.X%, X.X%) |
| Worse (Recanalization) | X.X% (n/N) | (X.X%, X.X%) |

Safety Analysis

| Primary Endpoint | | |
|---|---|---|
| | All Subjects (N = | |
| Safety Analysis | N) | 95% CI |
| | | (X.X%, |
| Procedural Device-Related Serious Adverse Events | X.X% (n/N) | X.X%) |

**Subject Deaths** 

| Subject Deaths | All Subjects (N = N) | 95% CI |
|---------------------|----------------------|--------------|
| One-Year Death Rate | X.X% (n/N) | (X.X%, X.X%) |

15

### **Serious Adverse Events**

| Serious Adverse Events | All Subjects (N = N) | 95% CI |
|------------------------|----------------------|--------------|
| Serious Adverse Events | X.X% (n/N) | (X.X%, X.X%) |
| SOC 1 | X.X% (n/N) | (X.X%, X.X%) |
| PT 1 | X.X% (n/N) | (X.X%, X.X%) |
| PT 2 | X.X% (n/N) | (X.X%, X.X%) |
| SOC 2 | X.X% (n/N) | (X.X%, X.X%) |
| PT 1 | X.X% (n/N) | (X.X%, X.X%) |
| PT 2 | X.X% (n/N) | (X.X%, X.X%) |

### **Device or Procedure Related Serious Adverse Events Within 24 hours**

| Device or Procedure Related Serious Adverse Events Within 24 hours Device or Procedure Related Serious Adverse Events All Subjects | | |
|---|---|---|
| Within 24 hours | (N = N) | 95% CI |
| | | (X.X%, |
| Device or Procedure Related Adverse Events | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| Device Related Adverse Events | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| SOC 1 | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| PT 1 | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| PT 2 | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| SOC 2 | X.X% (n/N) | X.X%) |
| | , , | (X.X%, |
| PT 1 | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| PT 2 | X.X% (n/N) | X.X%) |
| ••• | | (X.X%, |
| Procedure Related Adverse Events | X.X% (n/N) | (X.X%) |
| Troopagio Holdida / Idvoloo Evolito | 7 | (X.X%, |
| SOC 1 | X.X% (n/N) | X.X%) |
| | () | (X.X%, |
| PT 1 | X.X% (n/N) | X.X%) |
| | , , | (X.X%, |
| PT 2 | X.X% (n/N) | X.X%) |
| | , , | , |
| 111 | | |

**Device or Procedure Related Serious Adverse Events Greater than 24 hours** 

| Device or Procedure Related Serious Adverse | All Subjects (N = | |
|---------------------------------------------|-------------------|--------|
| Events Greater than 24 hours | N) | 95% CI |
| | | (X.X%, |
| Device or Procedure Related Adverse Events | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| Device Related Adverse Events | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| SOC 1 | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| PT 1 | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| PT 2 | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| Procedure Related Adverse Events | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| SOC 1 | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| PT 1 | X.X% (n/N) | X.X%) |
| | | (X.X%, |
| PT 2 | X.X% (n/N) | X.X%) |

**Subgroup Analysis: Actual Adjunctive Treatment Used** 

| Subgroup<br>Analysis | Balloon | 95% CI | Stent | 95% CI | Other | 95% CI | None | 95%<br>CI | P-<br>Value |
|---|---|---|---|---|---|---|---|---|---|
| Retreatment<br>through Follow-<br>Up | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.XXX |
| Adequate Occlusion at Immediate Post-Procedure | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.XXX |
| Re-Access<br>Attempts with<br>Guidewire due<br>to Catheter<br>Kickout | | | | | | | | | |
| 0 | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.XXX |
| 1 | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.XXX |
| 2 | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.XXX |
| ≥ 3 | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.X%<br>(n/N) | (X.X%,<br>X.X%) | X.XXX |

**Pooling Across Centers** 

| Pooli<br>ng<br>Acros<br>s<br>Cente<br>rs | Adjunctive<br>Treatment Used<br>(Yes/No) | Age ≥<br>65 | Aneury<br>sm<br>Locatio<br>n: ICA | Aneurysm<br>Size: Small | Aneurysm<br>Status:<br>Ruptured | Lesion<br>Nature:<br>Aneurysm | Lesion<br>Treatment<br>Technique<br>:<br>Deonstruct<br>ive | Neck<br>Width:<br>Wide<br>neck | Vessel<br>Treatment<br>at<br>Admission<br>:<br>Retreatme<br>nt |
|---|---|---|---|---|---|---|---|---|---|
| 99999 | X.X% (n/N) | X.X%<br>(n/N) | X.X%<br>(n/N) | X.X% (n/N) | X.X% (n/N) | X.X% (n/N) | X.X% (n/N) | X.X%<br>(n/N) | X.X% (n/N) |
| 99999 | X.X% (n/N) | X.X%<br>(n/N) | X.X%<br>(n/N) | X.X% (n/N)X | X.X% (n/N) | X.X% (n/N) | X.X% (n/N) | X.X%<br>(n/N) | X.X% (n/N) |
| P-<br>value | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |

**Major and Minor Protocol Deviations** 

| Major and Minor Protocol Deviations | All Subjects (N = N) |
|---|---|
| Major Deviations | |
| Subject does not Meet Inclusion Criteria | X.X% (n/N) |
| Subject was not Treated for Intracranial Aneurysms/ Other | |
| Neurovascular Abnormalities according to the Cleared | |
| Indications for SMART/PC 400/POD | X.X% (n/N) |
| Informed Consent not Obtained | X.X% (n/N) |
| Subject Meets Exclusion Criteria | X.X% (n/N) |
| Minor Deviations | |
| Improperly Signed or Incomplete Informed Consent | X.X% (n/N) |
| Out of Window Visit | X.X% (n/N) |
| Missing Visit | X.X% (n/N) |
| Out of Window Assessment | X.X% (n/N) |
| Assessment Not Done | X.X% (n/N) |
| Delayed Reporting of Serious or Procedure/Device Related | |
| Adverse Event | X.X% (n/N) |
| Registry Assessment/Procedure Done by Non Registry Staff or | |
| Registry Staff not Delegated to Task | X.X% (n/N) |
| Other | X.X% (n/N) |

**Enrollment and Screening** 

| Enrollment and Screening | All Subjects (N = N) |
|---|---|
| Consented and Not Enrolled | X.X% (n/N) |
| Less than 75% of Total Number of Coils Implanted are | |
| SMART, PC 400, or POD | X.X% (n/N) |
| Other | X.X% (n/N) |
| Not Consented and Not Enrolled | X.X% (n/N) |
| Did not Want to Participate | X.X% (n/N) |
| Life Expectancy less than 1 Year | X.X% (n/N) |
| Subject Already Enrolled in SMART | X.X% (n/N) |
| Participating in Another Clinical Investigation that could | |
| Confound the Evaluation of the Registry Device | X.X% (n/N) |
| Other | X.X% (n/N) |

**Sensitivity Analysis** 

| Sensitivity Analysis | All Subjects (N = N) | 95% CI |
|---|---|---|
| Analysis of All Subjects with Follow-Up | | |
| Complete | | |
| Retreatment through Follow-Up | X.X% (n/N) | (X.X%, X.X%) |
| Adequate Occlusion at Immediate Post- | | (X.X%, X.X%) |
| Procedure | X.X% (n/N) | |
| Re-Access Attempts with Guidewire due to | | |
| Catheter Kickout (SMART/PC 400/POD) | | |
| 0 | X.X% (n/N) | (X.X%, X.X%) |
| 1 | X.X% (n/N) | (X.X%, X.X%) |
| 2 | X.X% (n/N) | (X.X%, X.X%) |
| ≥ 3 | X.X% (n/N) | (X.X%, X.X%) |
| Procedural Device-Related Serious Adverse | | (X.X%, X.X%) |
| Events | X.X% (n/N) | , |
| Analysis of Complete Datasets with Missing | | |
| Data Imputed | | |
| Retreatment through Follow-Up | X.X% (n/N) | (X.X%, X.X%) |
| Adequate Occlusion at Immediate Post- | | (X.X%, X.X%) |
| Procedure | X.X% (n/N) | |
| Re-Access Attempts with Guidewire due to | | |
| Catheter Kickout (SMART/PC 400/POD) | X.X% (n/N) | |
| 0 | X.X% (n/N) | (X.X%, X.X%) |
| 1 | X.X% (n/N) | (X.X%, X.X%) |
| 2 | X.X% (n/N) | (X.X%, X.X%) |
| ≥ 3 | X.X% (n/N) | (X.X%, X.X%) |
| Procedural Device-Related Serious Adverse | , , | (X.X%, X.X%) |
| Events | X.X% (n/N) | , |

# Part II. Mock Listings

**Subject Follow-Up Visits** 

| Subject | Visit | Visit Date |
|-----------|----------------------|------------|
| | Admission Evaluation | |
| 99999-999 | Follow-Up | DDMONYYYY |

**Analysis Populations** 

| Subject | Intent-to-Treat | Per Protocol |
|-----------|-----------------|--------------|
| 99999-999 | Yes | Yes |
| | No | No |

**Subject Disposition** 

| Subject | Completed | If Yes, Date of<br>Registry<br>Completion | If No, Reason | Other,<br>Specify |
|---|---|---|---|---|
| 99999-999 | Yes<br>No | DDMONYYYY | Adverse Events Deceased before Completion Excluded for Medical Reasons Excluded from Registry by Investigator Lost to Follow Up Withdrew Consent Other | <specify text=""></specify> |

Demographics

| Subject | Age | Gender |
|-----------|-----|--------|
| 99999-999 | X | Female |
| | | Male |

**Medical History** 

| Subject | Medical History |
|-----------|----------------------------------------------|
| 99999-999 | Previous Stroke |
| | Headache |
| | Migraine |
| | Traumatic Brain Injury |
| | Myocardial Infarction |
| | Hypertension |
| | Thyroid Disorder |
| | Diabetes |
| | Other Past Medical History |
| | Family History of Aneurysms or Malformations |
| | Polycystic Kidney Disease |
| | Fibromuscular Dysplasia |
| | Smoking |
| | Cocaine Use |

#### **Process Times**

| | - | | Time from Arterial<br>Puncture to Last<br>Coil Detached |
|---|---|---|---|
| Subject | (Minutes) | (Minutes) | (Minutes) |
| 99999-999 | X | X | X |

#### **Lesion Evaluation**

| Subject | Technique | Previous<br>Treatment<br>with Coils | Lesion<br>Nature | Other,<br>Specify | Lesion<br>Side | Lesion<br>Locatio<br>n | Other,<br>Specify | Arterial<br>Access<br>Site | Other,<br>Specif<br>y |
|---|---|---|---|---|---|---|---|---|---|
| 99999-999 | Constructive<br>Deconstructive | Yes<br>No | Aneurysm<br>Fistula<br>Arterioven<br>ous<br>Malformati<br>on<br>Other | <specif<br>y text&gt;</specif<br> | Right<br>Left<br>Midline | Extradu ral ICA ICA ACA MCA Posterio r Circulati on Venous Circulati on Other | <specif<br>y text&gt;</specif<br> | Right Femoral Left Femoral Right Radial Left Radial Other, Specify | <speci<br>fy<br/>text&gt;</speci<br> |

**Adjunctive Treatment** 

| Subject | Adjunctive<br>Technology<br>Pre-<br>Planned | Planned Adjunctive<br>Treatment | Adjunctive<br>Technology<br>Used | Actual<br>Adjunctive<br>Treatment |
|---|---|---|---|---|
| 99999-999 | Yes<br>No | Stent-Assisted Coiling<br>Balloon-Assisted<br>Coiling<br>Other | Yes<br>No | Stent-Assisted Coiling Balloon-Assisted Coiling Other |

#### **Modified Rankin Scale**

| Subject | Admission mRS | One-Year mRS |
|-----------|---------------|--------------|
| 99999-999 | X | X |

**Hunt and Hess Grading Scale** 

| Subject | Admission Hunt and Hess |
|-----------|-------------------------|
| 99999-999 | X |

**Primary Effectiveness Analysis** 

| Subject | Retreatment through Follow-Up |
|-----------|-------------------------------|
| 99999-999 | Yes |
| | No |
| | Unknown |

**Secondary Effectiveness Analysis** 

| Subject | Was<br>Adequate<br>Occlusion<br>Achieved? | Occlusion of the | Re-Access<br>with<br>Guidewire<br>due to<br>Catheter<br>Kickout<br>while<br>Using<br>SMART/PC<br>400/POD | Re-Access<br>with<br>Guidewire<br>due to<br>Catheter<br>Kickout<br>while<br>Using<br>Other<br>Adjunctive | First Framing Coil<br>Conformed to<br>Lesion | Packing<br>Density | Occlusion<br>of the<br>Aneurysm<br>at One<br>Year | Occlusion<br>Grading of<br>Lesion at One<br>Year (Non- |
|---|---|---|---|---|---|---|---|---|
| Subject | Yes | Aneurysm<br>Not | 400/POD | Coils | Morphology | Density | rear | Aneurysm) |
| | No | Applicable | | | | | | |
| | | (no | | | | | | Better |
| | | aneurysm | | | | | Not | (Progressive |
| | | treated) | | | | | Applicable | Occlusion) |
| | | Class I<br>Class II | | | Completely | | (no<br>aneurysm | Stable<br>Worse |
| | | Class III | | | Conformed | | treated) | (Recanalization) |
| 99999-999 | | Not done, | Yes | Yes | Partially | X% | Class I | Not Applicable |
| | | explain: | No | No | Conformed | | Class II | (aneurysm |
| | | | | N/A | Compartmentalized | | Class III | treated) |
| i | | | | | N/A | | Not done, | Not done, |
| | | | I | | | | explain: | explain: |

Safety Analysis

| Subject Eve nt Date of Onset Continui ng) | Carety | | 70.0 | | | 1 | 1 | 1 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Nam e of Eve Date of Outcom e of Eve nt Onset Date Resolved Or Other, Specify | | | | | | | | | Balada | | |
| Nam e of Eve Date of Outcom nt | | / 17 | ĺ | Perioa | | | | | | ĺ | |
| Bubject Date of Conset Date of Outcom Procedure Subject Intraproced Unal or Within 24 Hours of Procedure After 24 Hours Procedure Proced | | / | | | | D-4- | | Dalatia malain ti | | | |
| Subject Eve nt Date of Onset Outcom e Or Other, Specify State/Angiogra phic Procedure POD Coil System Taken Specify State/Angiogra phic Procedure Pod Coil System State/Angiogra phic Procedure Pod Coil System Pod Coil Sys | | | | | | | | | | | 041 |
| Subject nt Onset e Specify y phic Procedure System Taken y Intraproced ural or within 24 hours of Procedure After 24 Hours Post Procedure this event Unresolv ed (Death Due to Other Event) Y or Specify Mild Probable Therapy fy | | | Data of | | 0 | | Carrania | | | Antina | Other, |
| Intraproced ural or within 24 ed (Event Procedure After 24 ng) Death due to this event Unresolv ed (Death Due to Other Event) Y or Specify Mild Probable Therapy fy | Cubicat | - | | | | , | | | | | Specif |
| ural or within 24 ed hours of Procedure After 24 Hours Post Procedure Unresolv ed (Death Due to Other Event) Unresolv ed (Death Due to Other Event) Unresolv especify Mild Probable Therapy fy | Subject | nτ | Unset | latas and and | | Specify | У | pnic Procedure | System | raken | У |
| within 24 hours of Procedure After 24 Hours Post Procedure Vert Procedure Pr | | | | | | | | | | | |
| hours of Procedure After 24 | | | | | | | | | | | |
| Procedure After 24 | | | | | | | | | | | |
| After 24 Hours Post Procedure After 24 Hours Post Procedure Death due to this event Unresolv ed (Death Due to Other Event) YY or Unresolv Specify Mild Unrelated Probable Remedial Frobable Therapy Fy | | | | | | | | | | | |
| Hours Post Procedure Hours Post Procedure Death due to this event Unresolv ed (Death Due to Other Event) YY or Possible Probable DDMONYY DDMONYY Hours Post Death due to this event Unresolv ed (Death Due to Other Event) YY or Possible Probable Therapy fy | | | | | | | | | | | |
| Procedure due to this event Unresolv ed (Death Due to Other Event) YY or Possible Remedial Specify Mild Probable Therapy fy | | | | | | | | | | | |
| this event Unresolv ed (Death Due to Other Event) YY or Possible Remedial Specify Mild Probable Therapy fy | | | | | | | | | | | |
| event Unresolv ed (Death Due to Other DDMONYY Event) YY or Possible Remedial Specify Mild Probable Therapy fy | | | | 1 Tocedure | | | | | | | |
| Unresolv ed (Death Due to Other DDMONYY Event) YY or Possible Remedial Specify Mild Probable Therapy fy | | | | | | | | | | | |
| ed (Death Due to Other DDMONYY Unrelated None Possible Remedial S Unresolv Specify Mild Probable Therapy fy | | | | | | | | | | | |
| (Death Due to Other DDMONYY Unrelated None Event) YY or Pobable Therapy fy | | | | | | | | | | | |
| Due to Other DDMONYY Unrelated None Remedial Specify Mild Probable Therapy fy | | | | | | | | | | | |
| Other Event) YY or Specify Mild Unrelated Possible Remedial Specify Mild Probable Therapy fy | | | | | | | | | | | |
| Seventy | | | | | | DDMONYY | | | Unrelated | None | |
| 99999- DDMONYY Unresolv Specify Mild Probable Therapy fy | | | | | - | | | | | | <speci< td=""></speci<> |
| ***** | 00000 | | DDMONVY | | | | Mild | | | | |
| | | Y | | | | | | Unrelated | | | text> |
| time of telephone Medical telephone we will be the possible N/A / Procedure | 333 | ^ | ' ' | | | ICAL> | | | | | ICAL- |
| registry Severe Probable Unrelated Hospitalizat | | | | | | | | | | | |
| l legistry Severe Probable Officialed Trospitalizat | | | | | | | Severe | | | | |
| y Unrelated Probable Other | | | ĺ | ĺ | | | | | | | |
| y officialed Probable Official Colorer Colorer Possible Definite | | | | | | | | | | Other | |
| Other Probable N/A / | | | | | | | | | | | |
| Definite Unrelated | | | | ĺ | Julion | | | | | | |
| Possible | | | ĺ | ĺ | | | | Domino | | ĺ | |
| Probable | | | | | | | | | | | |
| Definite | | | | | | | | | | | |

**Subject Deaths** 

| Subject | Date of Death |
|-----------|---------------|
| 99999-999 | DDMONYYYY |

#### **Serious Adverse Events**

| Seriou | 12 M | iverse E | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subje<br>ct | SO<br>C /<br>PT<br>/<br>Na<br>me<br>of<br>Eve<br>nt | Date of<br>Onset | Time<br>Period | Outco<br>me | Date<br>Resolve<br>d or<br>Other,<br>Specify | Sever<br>ity | Relationshi<br>p to Disease<br>State/Angio<br>graphic<br>Procedure | Relatio<br>nship to<br>SMART<br>/ PC 400<br>/ POD<br>Coil<br>System | Action<br>Taken | Othe<br>r,<br>Spec<br>ify | Classific<br>ation of<br>Event | Did<br>event<br>cause<br>the<br>subje<br>ct to<br>withd<br>raw<br>from<br>regist<br>ry? |
| 99999-999 | X | DDMON<br>YYYY | Intraproc<br>edural or<br>within 24<br>hours of<br>Procedur<br>e<br>After 24<br>Hours<br>Post<br>Procedur<br>e | Resolv ed Unreso lved (Event Contin uing) Death due to this event Unreso lved (Death Due to Other Event) Unreso lved (at time of registry exit/stu dy closure) Other | DDMON<br>YYYY or<br><specify<br>text&gt;</specify<br> | Mild<br>Mode<br>rate<br>Sever<br>e | Unrelated<br>Possible<br>Probable<br>Definite /<br>Unrelated<br>Possible<br>Probable<br>Definite | Unrelate d Possible Probabl e Definite / Unrelate d Possible Probabl e Unrelate d Possible Probabl e Definite / | None<br>Remedial<br>Therapy<br>Medical<br>Procedur<br>e<br>Hospitali<br>zation<br>Other | <spe<br>cify<br/>text&gt;</spe<br> | Death Permane nt impairme nt or damage Requires hospitaliz ation or prolongat ion of existing hospitaliz ation Life threateni ng Medical or surgical impairme nt to prevent permane nt impairme nt or damage | Yes<br>No |

### **Device or Procedure Related Adverse Events Within 24 hours**

| | SOC<br>/ PT<br>/<br>Nam<br>e of<br>Eve | Date of | Time<br>Period | Outcom | Date<br>Resolved<br>or Other, | Severit | Relationship to<br>Disease<br>State/Angiogra | Relations<br>hip to<br>SMART /<br>PC 400 /<br>POD Coil | Action | Other,<br>Specif |
|---|---|---|---|---|---|---|---|---|---|---|
| 99999-999 | X | DDMONYY<br>YY | Intraproced<br>ural or<br>within 24<br>hours of<br>Procedure<br>After 24<br>Hours Post<br>Procedure | Resolve d Unresolv ed (Event Continui ng) Death due to this event Unresolv ed (Death Due to Other Event) Unresolv ed (at time of registry exit/stud y closure) Other | DDMONYY YY or <specify text=""></specify> | Mild<br>Moder<br>ate<br>Severe | Unrelated Possible Probable Definite / Unrelated Possible Probable Definite | Unrelated Possible Probable Definite / Unrelated Possible Probable Definite / Unrelated Possible Definite / Unrelated Possible | None<br>Remedial<br>Therapy<br>Medical<br>Procedure<br>Hospitalizat<br>ion<br>Other | <speci<br>fy<br/>text&gt;</speci<br> |

#### **Device or Procedure Related Adverse Events Greater than 24 hours**

| Subject | SOC<br>/ PT<br>/<br>Nam<br>e of<br>Eve<br>nt | Date of<br>Onset | Time<br>Period | Outcom<br>e | Date<br>Resolved<br>or Other,<br>Specify | Severit<br>y | Relationship to<br>Disease<br>State/Angiogra<br>phic Procedure | Relations<br>hip to<br>SMART /<br>PC 400 /<br>POD Coil<br>System | Action<br>Taken | Other,<br>Specif<br>Y |
|---|---|---|---|---|---|---|---|---|---|---|
| 99999-999 | X | DDMONYY<br>YY | Intraproced<br>ural or<br>within 24<br>hours of<br>Procedure<br>After 24<br>Hours Post<br>Procedure | Resolve d Unresolv ed (Event Continuing) Death due to this event Unresolv ed (Death Due to Other Event) Unresolv ed (at time of registry exit/stud y closure) Other | DDMONYY<br>YY or<br><specify<br>text&gt;</specify<br> | Mild<br>Moder<br>ate<br>Severe | Unrelated<br>Possible<br>Probable<br>Definite /<br>Unrelated<br>Possible<br>Probable<br>Definite | Unrelated<br>Possible<br>Probable<br>Definite /<br>Unrelated<br>Possible<br>Probable<br>Definite /<br>Unrelated<br>Possible<br>Probable<br>Definite | None<br>Remedial<br>Therapy<br>Medical<br>Procedure<br>Hospitalizat<br>ion<br>Other | <speci<br>fy<br/>text&gt;</speci<br> |

**Enrollment and Screening** 

| | | | Reason<br>Subject<br>Not<br>Enrolled | Other,<br>Specify | Not<br>Consented<br>and Not<br>Enrolled | |
|---|---|---|---|---|---|---|
| Subject | Status | Date of Consent | Elifolieu | | Reason | Other, Specify |
| ousjeet | otacus | Date of Consont | Less than<br>75% of<br>total<br>number<br>of coils<br>implanted<br>are<br>SMART,<br>PC 400,<br>or POD<br>Other,<br>Specify | <specify<br>text&gt;</specify<br> | Did not want<br>to<br>participate<br>Life<br>expectancy<br>less than 1<br>year<br>Subject<br>already<br>enrolled in<br>SMART<br>Participating<br>in another | outer, opeany |
| Subject not<br>Consented | Consented<br>and Enrolled<br>Consented<br>and Not<br>Enrolled<br>Not<br>Consented<br>and Not<br>Enrolled | DDMONYYYY | | | clinical investigation that could confound the evaluation of the registry device Other | <specify text=""></specify> |

**Major and Minor Protocol Deviations** 

| Subject | Timepoint | Protocol Deviation Codes | Inclusion-Exclusion Criteria Not Met | Other,<br>Specify |
|---|---|---|---|---|
| 99999-999 | Baseline/Procedure<br>Discharge<br>Follow Up<br>Other (specify): | Subject does not Meet Inclusion Criteria Subject Meets Exclusion Criteria Improperly Signed or Incomplete Informed Consent Out of Window Visit Missing Visit Out of Window Assessment Assessment Not Done Delayed Reporting of Serious or Procedure/Device Related Adverse Event Registry Assessment/Procedure Done by Non Registry Staff or Registry Staff not Delegated to Task Other (specify): | Patient was not treated for intracranial aneurysms/ other neurovascular abnormalities according to the cleared indications for SMART/PC 400/ POD Informed consent not obtained Life expectancy is less than one year Participation in another clinical investigation that could confound the evaluation of the registry device Subject already enrolled in SMART registry | <specify text=""></specify> |

Part III. Mock Figures

Kaplan-Meier Estimates of Probability of Death in Subjects